CLINICAL TRIAL: NCT03254537
Title: Effect of Mediterranean Diets Based on Organic and Conventional Foods on Health Related Physiological Parameters in Urine and Blood/Plasma
Brief Title: Effect of Mediterranean Diets Based on Organic and Conventional Foods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Newcastle University (Other)
Collaborators: The Sheepdrove Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NUHEALTH-CS01-ORGANIC
Record Dates: First submitted 2017-06-21; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Health Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Organic (Experimental)
  Interventions: Dietary Supplement: Mediterranean Organic
- Mediterranean conventional (Experimental)
  Interventions: Dietary Supplement: Mediterranean conventional

INTERVENTIONS:
Dietary Supplement: Mediterranean Organic — Traditional Mediterranean diet comprised of organic ingredients
  Arms: Mediterranean Organic
Dietary Supplement: Mediterranean conventional — Traditional Mediterranean diet comprised of conventional ingredients
  Arms: Mediterranean conventional

SUMMARY:
Results from a small number of human cohort studies are also available and indicate that there are positive associations between organic food consumption and reduced risk/incidence of certain acute diseases (e.g. pre-eclampsia, hypospadias) and obesity/overweight.

Results from animal dietary intervention studies suggest that (i) switching to organic food consumption results in significant changes in hormonal balances and an increase in immune system responsiveness and (ii) differences in pesticide residue, cadmium, protein and antioxidant concentrations between organic and conventional foods are major drivers for hormonal balances and immune system parameters in animals.

However, there is virtually no published data from (i) long-term cohort studies focusing on chronic diseases (e.g. cardiovascular disease, diabetes, cancer and neurodegenerative conditions) and (ii) controlled human dietary intervention studies comparing effects of organic and conventional diets. It is therefore currently not possible to assess whether and estimate to what extent organic food consumption may affect human health.

DETAILED DESCRIPTION:
The most recent systematic literature reviews and meta-analyses have indicated significant and nutritionally-relevant composition differences between organic and conventional foods (crops, meat and dairy products). Specifically, these systematic reviews reported that:

organic crops have 17% higher antioxidant activity and between 18% and 69% higher concentrations of a range of individual antioxidants; increased intakes of polyphenolics and antioxidants has been linked to a reduced risk of certain chronic diseases such as cardiovascular and neurodegenerative diseases and certain cancers.

conventional crops have 48% higher levels of the toxic metal cadmium, and are 4-times more likely to contain detectable pesticide residues; there are general recommendations to minimise the intake of pesticides and cadmium to avoid potential negative health impacts.

conventional crops also have 15%, 10%, 30%, and 87% higher concentrations of protein, nitrogen, nitrate, nitrite, respectively; increased intakes of these compounds have been linked to both positive and negative health impacts.

organic meat, milk and dairy products have approximately 50% higher concentrations of nutritionally-desirable omega-3 fatty acids; intakes of very long chain omega-3 fatty acids in Western diets and there are EFSA recommendation to at least double their intake.

organic milk has 70% lower concentrations of iodine and slightly lower concentrations of Selenium, which is nutritionally undesirables especially in the UK where (a) the Se content of cereals has decreased (due to reduced import of cereals grown on Se-rich soil (b) Iodine fortified table salt is not widely available and used and the iodine supply relies more on mineral fortification of animal, and especially dairy feeds.

Results from a small number of human cohort studies are also available and indicate that there are positive associations between organic food consumption and reduced risk/incidence of certain acute diseases (e.g. pre-eclampsia, hypospadias) and obesity/overweight .

Results from animal dietary intervention studies suggest that (i) switching to organic food consumption results in significant changes in hormonal balances and an increase in immune system responsiveness and (ii) differences in pesticide residue, cadmium, protein and antioxidant concentrations between organic and conventional foods are major drivers for hormonal balances and immune system parameters in animals.

However, there is virtually no published data from (i) long-term cohort studies focusing on chronic diseases (e.g. cardiovascular disease, diabetes, cancer and neurodegenerative conditions) and (ii) controlled human dietary intervention studies comparing effects of organic and conventional diets. It is therefore currently not possible to assess whether and estimate to what extent organic food consumption may affect human health.

The overall aim of the study is to get a quantitative understanding of (a) the uptake (and therefore potential to affect health) of food composition components (pesticide residues, toxic metals such as cadmium, antioxidants) that differ between organic and conventional foods and (b) the effect of organic vs conventional food consumption on selected physiological parameters in plasma linked to health.

This information will be essential to (a) carry out accurate statistical power analyses (based on uptake [=estimated from blood and urine concentrations] rather than food composition data) and (b) optimise designs for longer-term dietary intervention studies, designed to identify impacts of organic food consumption on health related physiological markers in humans and mechanisms for potential health impacts.

The main objectives of the proposed study are to:

1. Carry out a human dietary intervention study comparing the effects of switching to Mediterranean diets based on organic and conventional foods on concentrations of pesticides, toxic metals, mineral nutrients (e.g. Fe, Cu, Se, I) and antioxidants, and antioxidant activity and selected health-related markers in urine and blood.
2. Quantify concentrations of pesticide residue, mineral, toxic metal and antioxidants in both organic and conventional food samples consumed during the intervention period
3. Carry out both univariate and redundancy analyses to both quantify effects of different diets on urine and blood composition and to identify the most important food composition drivers for differences in urine/blood composition and health markers.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults No medications No known illness

Exclusion Criteria:

Any known illness Using prescribed medication Using over the counter vitamin or mineral supplements Allergy to any food

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
IL-6 in Plasma measured using ELISA | Change from baseline 2 weeks post supplementation and 4 weeks post supplementation
IL-6 in WBC measured using ELISA | Change from baseline 2 weeks post supplementation and 4 weeks post supplementation
DNA damage in WBC measured using Western Blot | Change from baseline 2 weeks post supplementation and 4 weeks post supplementation
Total antioxidant activity in plasma measured using PENTRA | Change from baseline 2 weeks post supplementation and 4 weeks post supplementation
Phenols in plasma measured using GCMS | Change from baseline 2 weeks post supplementation and 4 weeks post supplementation
Carotenoids in plasma measured using GCMS | Change from baseline 2 weeks post supplementation and 4 weeks post supplementation
Pesticides in urine and plasma measured using ICPMS | Change from baseline 2 weeks post supplementation and 4 weeks post supplementation
Isoprostanes in urine measured using ICPMS | Change from baseline 2 weeks post supplementation and 4 weeks post supplementation
toxic metals in urine and plasma (Cd, Pb, Hg, Al) measured using ICPMS | Change from baseline 2 weeks post supplementation and 4 weeks post supplementation
minerals in plasma (including Cu, Fe, Mn, Mg, Ca, I, Se) measured using ICPMS | Change from baseline 2 weeks post supplementation and 4 weeks post supplementation

CONTACTS AND LOCATIONS:
Locations (2):
- Levidopa Field Station, Sivas, Sivas Festos, Greece
- NU-Food Research Facility, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rempelos L, Wang J, Baranski M, Watson A, Volakakis N, Hadall C, Hasanaliyeva G, Chatzidimitriou E, Magistrali A, Davis H, Vigar V, Srednicka-Tober D, Rushton S, Rosnes KS, Iversen PO, Seal CJ, Leifert C. Diet, but not food type, significantly affects micronutrient and toxic metal profiles in urine and/or plasma; a randomized, controlled intervention trial. Am J Clin Nutr. 2022 Nov;116(5):1278-1290. doi: 10.1093/ajcn/nqac233. Epub 2023 Feb 10. PMID 36041176
- [Derived] Rempelos L, Wang J, Baranski M, Watson A, Volakakis N, Hoppe HW, Kuhn-Velten WN, Hadall C, Hasanaliyeva G, Chatzidimitriou E, Magistrali A, Davis H, Vigar V, Srednicka-Tober D, Rushton S, Iversen PO, Seal CJ, Leifert C. Diet and food type affect urinary pesticide residue excretion profiles in healthy individuals: results of a randomized controlled dietary intervention trial. Am J Clin Nutr. 2022 Feb 9;115(2):364-377. doi: 10.1093/ajcn/nqab308. PMID 34718382